CLINICAL TRIAL: NCT03946995
Title: Comparison of Dry Needling and Graston Technique in Active Myofascial Trigger Points on Upper Trapezius
Brief Title: Dry Needling Versus Graston Technique in Active Myofascial Trigger Points on Upper Trapezius
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: RiphahIU Kiran Haq
Record Dates: First submitted 2019-05-09; First posted 2019-05-13 (Actual); Last update posted 2019-08-09 (Actual); Status verified 2019-08

CONDITIONS: Trigger Points
Keywords: Trigger Area; Myofascial Pain Syndromes; Instrument assisted soft tissue tecnique
MeSH Terms: conditions — Myofascial Pain Syndromes

STUDY DESIGN:
Intervention Model Description: There will be two treatment groups of participants, One group will receive Dry Needling whereas other will receive Graston technique for treatment of Myofascial Trigger points.
Who Masked: Participant
Masking Description: This is a single blinded randomized controlled trial in which patients will be randomized into groups by sealed envelope method.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dry needling (Experimental): Dry needling will be applied on active myofascial trigger points in upper trapezius along with conservative physical therapy management.
  Interventions: Other: Dry Needling Group
- Graston (Active Comparator): Graston Technique will be applied on active myofascial trigger points in upper trapezius along with conservative physical therapy management.
  Interventions: Other: Graston Technique Group

INTERVENTIONS:
Other: Dry Needling Group — Hot Pack will be applied on upper trapezius muscles before session for general relaxation for 7-10 minutes. Generalized Stretching and strengthening neck exercises will be performed. Then after wearing gloves and appropriate personal protective measures, a thin filiform needle will be inserted which will penetrate into the skin and stimulate underlying myofascial trigger points.
  The treatment will be continued for 2 weeks with 2 sessions per week.
  Arms: Dry needling
Other: Graston Technique Group — Hot Pack will be applied on upper trapezius muscles before session for general relaxation for 7-10 minutes. Generalized Stretching and strengthening neck exercises will be performed.
  Later, lubricant will be applied to the skin, and Graston technique will be applied using instrument over the active myofascial trigger points in upper trapezius.
  The treatment will be continued for 2 weeks with 2 sessions per week.
  Arms: Graston

SUMMARY:
This study will compare the effects dry needling and Graston technique in active myofascial trigger points on upper trapezius. Half of the study participants will receive dry needling whereas other half will receive Graston technique.

DETAILED DESCRIPTION:
This is a single blinded randomized controlled trial, will be conducted at Rawal General & Dental Hospital, Islamabad. Both dry needling and Graston Techniques are used to release active Myofascial Trigger points with different mechanism.

Dry needling is technique in which without any medication or injection, dry needles are inserted into hyper irritable points in muscle. Graston technique is done with specially designed tools to locate knots within muscle by running the tools over the skin.

This study is planned with objectives to compare both treatment techniques on active myofascial trigger points in patients with neck pain. Effects of these will be measured on Neck Pain, Range of Motion, functional status and trigger points.

ELIGIBILITY:
Inclusion Criteria:

* Patient with non-specific pain in neck (acute and sub-acute)
* Age: 20-40 years
* Patient agrees to use the dry needling or Graston exclusively

Exclusion Criteria:

* Patients that were using any medication to reduce the pain and/or have any effect in the skeleton muscle.
* Patient taking other treatment in the same period of research.
* Patients having malignancy, tuberculosis, spinal cord injury, neurodegenerative diseases radiculopathies and hematoma.
* Patients on anticoagulants.
* Patient with chronic neck pain.

Ages: 20 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2019-03-19 (Actual); Primary Completion 2019-06-30 (Actual); Study Completion 2019-06-30 (Actual)

PRIMARY OUTCOMES:
Numeric Pain Rating Scale (NPRS) | Baseline
  Numeric Pain Rating Scale (NPRS) is used to assess pain. It scores ranges from 0-10, 0 means No pain and 10 means Severe pain. Patient will be asked to verbally report the pain score.
Numeric Pain Rating Scale (NPRS) | Post 2nd week
  Numeric Pain Rating Scale (NPRS) is used to assess pain. It scores ranges from 0-10, 0 means No pain and 10 means Severe pain. Patient will be asked to verbally report the pain score.
cervical range of motion (CROM) | Baseline
  A cervical range of motion (CROM) inclinometer will be use to assess cervical range of motion in flexion, extension, left right lateral flexion and left-right rotation. Participants will be seated upright and asked to actively move their neck in each direction.
cervical range of motion (CROM) | Post 2nd week
  A cervical range of motion (CROM) inclinometer will be use to assess cervical range of motion in flexion, extension, left right lateral flexion and left-right rotation. Participants will be seated upright and asked to actively move their neck in each direction.
Myofascial Diagnostic Scale (MDS) | Baseline
  It is a scale using the signs of a Myofascial trigger point as indicators to assess the extent to which the patient suffers from Myofascial Pain Syndrome.
  The signs include: referred pain in the zone of reference, local twitch response, palpable taut band, and focal or spot tenderness.
  Spot tenderness or soft tissue tenderness consisted of five grades or indicators: grade 0 - no tenderness = 0, grade 1 - tenderness to palpation without grimace or flinch = 1, grade 2 - tenderness with grimace and/or flinch to palpation = 2, grade 3 - tenderness with withdrawal = 3, grade 4 - withdrawal to non-noxious stimuli = 4.
  The presence of a local twitch response and the presence of a palpable taut band were indicated by a score of 4 on the scale.
  The presence of referred pain was indicated by a score of 5. A total score of 9 or more was indicative of active trigger points.
Myofascial Diagnostic Scale (MDS) | Post 2nd Week
  It is a scale using the signs of a Myofascial trigger point as indicators to assess the extent to which the patient suffers from Myofascial Pain Syndrome.
  The signs include: referred pain in the zone of reference, local twitch response, palpable taut band, and focal or spot tenderness.
  Spot tenderness or soft tissue tenderness consisted of five grades or indicators: grade 0 - no tenderness = 0, grade 1 - tenderness to palpation without grimace or flinch = 1, grade 2 - tenderness with grimace and/or flinch to palpation = 2, grade 3 - tenderness with withdrawal = 3, grade 4 - withdrawal to non-noxious stimuli = 4.
  The presence of a local twitch response and the presence of a palpable taut band were indicated by a score of 4 on the scale.
  The presence of referred pain was indicated by a score of 5. A total score of 9 or more was indicative of active trigger points.

SECONDARY OUTCOMES:
Neck Disability Index (NDI) | Baseline
  Neck Disability Index (NDI) is a questionnaire designed to assess how neck pain has affected patient's ability to manage in everyday life. It has total 10 sections, For each section the total possible score is 5: if the first statement is marked the section score = 0, if the last statement is marked it = 5. If all ten sections are completed the score is calculated and converted into percentages. The maximum Score of Neck Disability Index (NDI) is 50.
Neck Disability Index (NDI) | Post 2nd week
  Neck Disability Index (NDI) is a questionnaire designed to assess how neck pain has affected patient's ability to manage in everyday life. It has total 10 sections, For each section the total possible score is 5: if the first statement is marked the section score = 0, if the last statement is marked it = 5. If all ten sections are completed the score is calculated and converted into percentages. The maximum Score of Neck Disability Index (NDI) is 50.

CONTACTS AND LOCATIONS:
Overall Officials: Huma Riaz, Principal Investigator — Riphah International University
Locations (1):
- Rawal General and Dental Hospital,, Islamabad, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gerber LH, Shah J, Rosenberger W, Armstrong K, Turo D, Otto P, Heimur J, Thaker N, Sikdar S. Dry Needling Alters Trigger Points in the Upper Trapezius Muscle and Reduces Pain in Subjects With Chronic Myofascial Pain. PM R. 2015 Jul;7(7):711-718. doi: 10.1016/j.pmrj.2015.01.020. Epub 2015 Feb 4. PMID 25661462
- [Background] Dunning J, Butts R, Mourad F, Young I, Flannagan S, Perreault T. Dry needling: a literature review with implications for clinical practice guidelines. Phys Ther Rev. 2014 Aug;19(4):252-265. doi: 10.1179/108331913X13844245102034. PMID 25143704
- [Background] Wang G, Gao Q, Hou J, Li J. Effects of Temperature on Chronic Trapezius Myofascial Pain Syndrome during Dry Needling Therapy. Evid Based Complement Alternat Med. 2014;2014:638268. doi: 10.1155/2014/638268. Epub 2014 Oct 14. PMID 25383083
- [Background] Gattie ER, Cleland JA, Snodgrass SJ. Dry Needling for Patients With Neck Pain: Protocol of a Randomized Clinical Trial. JMIR Res Protoc. 2017 Nov 22;6(11):e227. doi: 10.2196/resprot.7980. PMID 29167092